CLINICAL TRIAL: NCT01095380
Title: Comparison of Post-SCI Locomotor Training Techniques
Brief Title: Comparison of Post-pinal Cord Injury (SCI) Locomotor Training Techniques
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Edelle Field-Fote, Professor, University of Miami Miller School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD041487 (NIH)
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2009-01

CONDITIONS: Spinal Cord Injury
Keywords: task-specific training; walking; locomotion; function; body weight support; Individuals with motor-incomplete spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treadmill training - manual assist (TM) (Active Comparator): Participants in the TM group received partial body weight support unilateral or bilateral manual assistance from a trainer for stepping
  Interventions: Other: Locomotor training
- Treadmill training - electrical stimulation (TS) (Active Comparator): Participants in the TS group received partial body weight support and bilateral functional electrical stimulation to assist stepping
  Interventions: Other: Locomotor training
- Overground Training (OG) (Active Comparator): Training over ground with body weight support and electrical stimulation for dorsiflex assistance
  Interventions: Other: Locomotor training
- Treadmill training - locomat robot (LR) (Active Comparator): Treadmill training with partical body weight support and assistance of a robotic gait orthosis for stepping
  Interventions: Other: Locomotor training

INTERVENTIONS:
Other: Locomotor training — Locomotor training using body weight support with training on a treadmill or training over ground with differing forms of assistance for stepping

SUMMARY:
Background: Body weight supported (BWS) locomotor training improves overground walking ability in individuals with motor-incomplete spinal cord injury (SCI). While there are various approaches available for locomotor training, there is no consensus regarding which of these is optimal. The purpose of this ongoing investigation is to compare outcomes associated with these different training approaches.

Subjects and Methods: Subjects with chronic motor-incomplete SCI have completed training and initial and final testing. Subjects were randomly assigned to 1 of 4 different BWS assisted-stepping groups, including: 1) treadmill training with manual assistance (TM), 2) treadmill training with stimulation (TS), 3) overground training with stimulation (OG), or 4) treadmill training with robotic assistance (LR). Prior to and following participation the investigators assessed:

* Walking-related outcome measures: overground walking speed, training speed, step length and step symmetry.
* Spinal cord reflex activity
* Electromyographic (EMG) associated with walking

Hypotheses:

In individuals with incomplete spinal cord injury (SCI):

1. A 12-week period of body weight supported treadmill training with TS will produce improvements in walking function that are significantly greater than those produced by training with TM, OG, LR.
2. TS training will be associated with greater changes to spinal reflex activity than will be observed in subjects trained with manual assistance or non-assisted stepping. Changes to spinal reflex activation will be such that this activity more closely resembles that observed in non-disabled (ND) individuals.
3. Following participation in this walking regimen, EMG activity observed during walking in all groups will be more robust, more consistent and better coordinated than EMG measures obtained prior to training.

ELIGIBILITY:
Inclusion Criteria:

* motor-incomplete spinal cord injury (AIS C or D)
* at least one year post injury
* able to step with at at least one leg
* able to stand from chair with no more than moderate assist of 1 person

Exclusion Criteria:

* unstable neurologic status
* active orthopedic problem

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2003-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Walking speed | 12 weeks
  Walking speed collected during 10-Meter Walk Test

SECONDARY OUTCOMES:
Functional walking capacity | 12 weeks
  Distance walked in timed 2-Minute Walk Test

CONTACTS AND LOCATIONS:
Overall Officials: Edelle C Field-Fote, PT, PhD, Principal Investigator — University of Miami

REFERENCES:
- [Result] Field-Fote EC, Lindley SD, Sherman AL. Locomotor training approaches for individuals with spinal cord injury: a preliminary report of walking-related outcomes. J Neurol Phys Ther. 2005 Sep;29(3):127-37. doi: 10.1097/01.npt.0000282245.31158.09. PMID 16398945
- [Result] Field-Fote EC, Brown KM, Lindley SD. Influence of posture and stimulus parameters on post-activation depression of the soleus H-reflex in individuals with chronic spinal cord injury. Neurosci Lett. 2006 Dec 13;410(1):37-41. doi: 10.1016/j.neulet.2006.09.058. Epub 2006 Oct 12. PMID 17046161
- [Result] Field-Fote EC, Dietz V. Single joint perturbation during gait: preserved compensatory response pattern in spinal cord injured subjects. Clin Neurophysiol. 2007 Jul;118(7):1607-16. doi: 10.1016/j.clinph.2007.03.022. Epub 2007 May 1. PMID 17475549
- [Result] Ness LL, Field-Fote EC. Whole-body vibration improves walking function in individuals with spinal cord injury: a pilot study. Gait Posture. 2009 Nov;30(4):436-40. doi: 10.1016/j.gaitpost.2009.06.016. Epub 2009 Aug 3. PMID 19648013
- [Result] Nooijen CF, Ter Hoeve N, Field-Fote EC. Gait quality is improved by locomotor training in individuals with SCI regardless of training approach. J Neuroeng Rehabil. 2009 Oct 2;6:36. doi: 10.1186/1743-0003-6-36. PMID 19799783
- [Derived] Sandler EB, Roach KE, Field-Fote EC. Dose-Response Outcomes Associated with Different Forms of Locomotor Training in Persons with Chronic Motor-Incomplete Spinal Cord Injury. J Neurotrauma. 2017 May 15;34(10):1903-1908. doi: 10.1089/neu.2016.4555. Epub 2017 Jan 4. PMID 27901413